



| IRAS ID: | R&D reference Number: | PEOS ID Number: | Participant Identification Number: |
|---|---|---|---|
| 286913 | 21/OPH/606 | 2669 | |

## **Participant Consent Form**

**Full Study title:** Vision and balance change after bilateral implantation of Toric versus non-Toric intraocular lenses in cataract patients with astigmatism.

| Chief Investigator: Prof Phillip Buckhurst | Principal Investigator: Prof Nabil Habib |
|---|---|
| Co - Investigators: Dr Catriona MacLennan, Prof Gary Shum, Dr Hetal Buckhurst, Ms Sherrie Choy | |

Please initial box if you agree with the accompanying statements below:

| | Statements | Initials: |
|---|---|---|
| , | . I confirm that I have read the participant information sheet (version 1.0 April 2022) for the above | |
| | study. | |
| 2 | . I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 3 | . I understand that my participation is voluntary and that I am free to withdraw at any time without | |
| | giving any reason, without my medical care or legal rights being affected. | |
| 2 | . I understand that if I withdraw from the study research data about me collected up to that point may be used by the research team, but the data will be anonymous and it will not be possible to identify me. | |
| ţ | . I understand that relevant sections of my medical notes and data collected during the study, may be looked at by the research team members named above, from the regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| 6 | . I understand that identifiable data about me will be shared between University Hospitals Plymouth | |
| | NHS Trust and the University of Plymouth. | |
| 7 | I understand that the information collected about me will be used to support<br>other research or education activities in the future and in this instance, my data would be<br>anonymous, and I would not be identifiable either directly or indirectly. | |
| 8 | . I understand that my data will be securely destroyed after 10 years of secure storage at University Hospitals Plymouth NHS Trust in accordance with Trust Policy. | |
| Ş | . I agree to my General Practitioner (GP) being informed of my participation in the study, and that they can be contacted to obtain relevant medical information about me if required. | |
| , | I agree to take part in the above study. | |

| Name of person giving consent (participant): | Researcher/ investigator name: |
|---|---|
| Signature of person giving consent (participant): | Researcher/ investigator Signature |
| Date: | Date |

<sup>\*1</sup>copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes.